CLINICAL TRIAL: NCT00117377
Title: Effects of Pimecrolimus Cream 1% on the Molecular and Cellular Profile of Adult Male Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981C2436
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, pimecrolimus, cellular, molecular
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus
- 2 (Placebo Comparator): Placebo control twice daily application
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 % bid
  Other Names: Elidel
  Arms: 1
Drug: Placebo — Placebo application bid
  Arms: 2

SUMMARY:
The purpose of this study is to identify how pimecrolimus cream 1% modifies the molecular and cellular changes associated with the post-lesional phase of atopic dermatitis (AD). Healthy volunteers and patients with atopic dermatitis will be studied.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with atopic dermatitis:

* Outpatient at screening
* Adult male >20 years old
* Diagnosis of AD fulfilling the Hannifin and Rajka criteria
* Mild to moderate AD (Investigator Global Assessment [IGA] 2-3; localized eczema area and severity index [EASI] 1-8)
* AD affecting both arms and/or legs >10cm2 per target area
* Willing to undergo 4 mm serial punch biopsies
* Patient history of AD for at least 3 years

Inclusion criteria for healthy volunteers:

* Volunteers must be males >20 years of age
* Volunteers must be in good health, as determined by past medical history, physical examination, and vital signs

Exclusion Criteria:

Exclusion criteria for patients with atopic dermatitis:

* Concurrent diseases/conditions and history of other diseases/conditions
* Are immunocompromised or have a history of malignant disease
* Have a history of rheumatic fever, heart valve replacement, prosthetic joints or other prosthetic constituents
* Have concurrent skin disease (e.g. acne) of such severity in the study area that it could interfere with the study evaluation
* Have previously reported poor or no clinical response to topical tacrolimus ointment (Protopic®) or pimecrolimus cream (Elidel®)
* Have active skin infections
* Present with clinical conditions other than atopic dermatitis that can interfere with the study treatment
* Present with severe medical condition(s) that, in the opinion of the investigator, prohibits participation in the study
* Are maintained on emollients that contain supplementary ingredients such as urea, alpha or beta-hydroxy acids, fruit acids, vitamins A, D or E
* Have received phototherapy (e.g. UVA, UVB) or systemic therapy (e.g. immunosuppressants, cytostatics) known or suspected to have an effect on AD within 4 weeks of Visit 1 (screening)
* Have received systemic corticosteroids ([CS] e.g. oral, intravenous, intraarticular, rectal) within 4 weeks of Visit 1 (screening). Patients on a stable maintenance dose of inhaled or intranasal CS may participate
* Were treated with topical therapy, including topical calcineurin inhibitors (e.g. corticosteroids, tar) known or suspected to have an effect on AD during the current acute episode
* Were treated with antihistamines within 7 days of Visit 1
* Known serious adverse reactions or hypersensitivity to anesthetics such as lidocaine or mepivacaine
* Excluded investigational drugs/hypersensitivity
* Have received investigational drugs within 8 weeks of the first application of study drug or planned use of other investigational drugs during participation in this study
* Have known hypersensitivity to any ingredient of the pimecrolimus cream 1% or this class of study drug

Exclusion criteria for healthy volunteers:

* Erythrodermic patients, patients with Netherton's syndrome
* Personal or family history of atopy (asthma, allergic rhinitis, atopic dermatitis)
* Clinically significant findings during the physical examination
* Have a history of rheumatic fever, heart valve replacement, prosthetic joints or other prosthetic constituents e.g. lens implants or hip joints
* Volunteers with known serious adverse reactions or hypersensitivity to anesthetics such as lidocaine or mepivacaine
* Participation in any clinical trial within one month prior to current trial
* History of immunocompromise
* History of positive hepatitis B surface antigen (HBsAg) or hepatitis C test result
* Use of corticosteroids within 4 weeks prior to baseline
* Were treated with antihistamines within 7 days of Visit 1
* Phototherapy within 4 weeks prior to baseline
* Topical therapy within 5 weeks prior to the study
* Treatment with nephrotoxic drugs within 2 weeks prior to baseline (aminoglycosides, amphotericin B, colchicine)

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-04; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Determining whether pimecrolimus cream has an effect on the cellular and molecular profile of atopic dermatitis skin, which is cleared of lesions and is otherwise clinically normal.

SECONDARY OUTCOMES:
Identifying cellular and molecular changes in skin in an acute phase of atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Mount Sinai School of Medicine, New York, New York
  - New York University Hospital, New York, New York
  - Virginia Clinical Research, Inc, Norfolk, Virginia